CLINICAL TRIAL: NCT00061269
Title: Videoendoscopic Drainage of Infected Pancreatic Collections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VDIPC (completed); R03DK061362 (NIH)
Record Dates: First submitted 2003-05-22; First posted 2003-05-23 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Pancreatitis, Acute Necrotizing
Keywords: Infected pancreatic necrosis
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VARD (Experimental): Videoscopic-Assisted Retroperitoneal Debridement (VARD)
  Interventions: Procedure: Videoscopic-Assisted Retroperitoneal Debridement (VARD)

INTERVENTIONS:
Procedure: Videoscopic-Assisted Retroperitoneal Debridement (VARD)

SUMMARY:
The VARD (Videoendoscopic Assisted Retroperitoneal Drainage) approach as treatment for necrotizing pancreatitis proposes an alternative to standard complicated open abdomen treatment methods.

This treatment involves making a small incision and looking inside the abdomen with a videoendoscope. A videoendoscope is an instrument with a small camera and light on the end. It also has an extension tool that the surgeon can use to clean out any dead and infected tissue in the abdomen.

This approach may reveal a treatment opportunity with faster recovery potential and shorter hospitalizations for patients with necrotizing pancreatitis.

ELIGIBILITY:
* Pancreatic necrosis or peripancreatic fluid collection following acute pancreatitis noted on CT scan
* Infected pancreatic necrosis or pancreatic abscess and determined by + FNA (gram stain or culture), as defined by the Atlanta Symposium
* Not neutropenic or pregnant
* No prior necrosectomy
* No pancreatic pseudocyst, either sterile or infected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-09 (Actual); Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Oregon Health Sciences University, Portland, Oregon
  - Veteran's Administration-Portland, Portland, Oregon
  - Harborview Medical Center, Seattle, Washington
  - Veteran's Administration Puget Sound, Seattle, Washington
  - University of Washington, Seattle, Washington
- University of Toronto, Toronto, Ontario, Canada